CLINICAL TRIAL: NCT02043535
Title: Effects of Controlled Hypercapnic Stimulation on Myocardial Blood Flow Measured With Positron Emission Tomography
Brief Title: CO2 as a Stress Agent for Perfusion Imaging
Acronym: CO2 STRESS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The complexity of the study and the recent slow down situation hampered the ability to recruit CAD patients therefore the study has been terminated.
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Terrence Ruddy, MD, Ottawa Heart Institute Research Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20140012
Record Dates: First submitted 2014-01-03; First posted 2014-01-23 (Estimated); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Coronary Artery Disease
Keywords: myocardial perfusion imaging; myocardial blood flow; pharmacologic stress agents; carbon dioxide; rubidium 82 radioisotope; positron emission tomography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Myocardial blood flow quantification (Other): The RA-MR™ Virtual Sequential Gas Delivery System. : delivery of CO2 in increasing levels.
  Rubidium Elution System: delivery of Rb-82 through an automated pump system for myocardial PET perfusion imaging.
  Persantine stress myocardial PET perfusion imaging: as a standard for comparison.
  Interventions: Device: Delivery of precise levels of carbon dioxide with the RA-MR™ Virtual Sequential Gas Delivery System.; Device: Delivery of rubidium radioisotope (Rb-82) using the automated pump/elution system

INTERVENTIONS:
Device: Delivery of precise levels of carbon dioxide with the RA-MR™ Virtual Sequential Gas Delivery System. — All participants will undergo a baseline rest Rb-82 positron emission tomography (PET) myocardial perfusion imaging scan (MPI) with low-dose computed tomography. Following this baseline study, serial Rb-82 PET MPI using a target level of carbon dioxide (CO2) (approximately 60 mmHg (± 3 mmHg)) as a stress agent will be performed. The 60 mmHg level will be repeated following a minimum 10 minute rest. A rest/stress Rb-82 PET MPI will be performed after return to normal CO2 levels (normocapnea) using persantine as the stress agent.
  Myocardial perfusion stress testing
  Other Names: the RA-MR™ System
Device: Delivery of rubidium radioisotope (Rb-82) using the automated pump/elution system — All participants will undergo a baseline rest Rb-82 positron emission tomography myocardial perfusion imaging scan (PET MPI) with low-dose CT. Following this baseline study, serial Rb-82 PET MPI using three target levels of pulmonary end-tidal carbon dioxide tension (PetCO2) (approximately 60 mmHg (± 3 mmHg)) as a stress agent will be performed. The 60 mmHg level will be repeated following a minimum 10 minute rest. A second rest Rb-82 PET MPI will be performed after return to normocapnea, followed by a pharmacologic persantine stress Rb-82 PET MPI.
  Other Names: Ruby-Fill™

SUMMARY:
Myocardial perfusion imaging (MPI) is a nuclear scan using a radioisotope to see blood flow to the muscles of the heart when the heart is at rest and when it is under stress. The stress test in MPI can be done using medications, such as persantine, that dilate coronary arteries and increase blood flow. Similarly, elevated carbon dioxide (CO2) levels in the blood, or hypercapnia, also dilates arteries and increases blood flow. Thornhill Research Inc. has developed the RA-MR™ sequential gas delivery system used to control CO2 levels in the blood. The RA-MR™ can deliver precise amounts of CO2 through a mouthpiece for inhalation to increase CO2 levels in the blood and thereby increasing blood flow like during stress.

The objective of this study is to compare the differences in blood flow through the arteries of the heart during stress with hypercapnia and adenosine MPI. The imaging will be done using positron emission tomography (PET) with the radioisotope, or tracer, called Rubidium (Rb-82). The Rb-82 is given through a pump, or elution system.

The investigators hypothesize that hypercapnia will induce a stress-to-rest increase in myocardial blood flow by a factor of 2 or more in myocardial regions supplied by non-stenotic arteries in normal volunteers and participants with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

For all participants

* Age ≥ 18 years old
* BMI ≤ 40 kg/m2
* Able and willing to comply with the study procedures
* Written informed consent
* Participants with documented coronary artery disease
* Stable coronary artery disease on a stable medication regime.
* Healthy volunteers without known heart disease
* Low risk of coronary artery disease (CAD)

Exclusion Criteria:

* History or risk of severe bradycardia (heart rate < 50 beats per minute) not related to chronotropic drugs
* Known second- or third-degree Atrio-ventricular block without pacemaker
* Atrial flutter or atrial fibrillation
* Dyspnea (NYHA III/IV), wheezing asthma or Chronic Obstructive Pulmonary Disease (COPD)
* Coronary artery bypass graft (CABG) surgery within 60 days prior to screening or at any time after consent
* Percutaneous coronary intervention (PCI) within 30 days prior to screening or at any time following consent
* Acute myocardial infarction or acute coronary syndrome within 60 days prior to screening or at any time following consent
* Recent use of dipyridamole, dipyridamole-containing medications (e.g. Aggrenox)
* Known hypersensitivity to adenosine
* Breastfeeding or pregnancy
* Claustrophobia or inability to lie still in a supine position
* Unwillingness or inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03-12 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Myocardial blood flow differences | Difference between baseline rest scan blood flow and hypercapnia stress scan myocardial blood flow at 50 mmHg, 55 mmHg, 60 mmHg levels from baseline. Imaging and intervention analysis will be complete in 4 years.
  The myocardial blood flow (MBF) will be quantified with each Rb-82 PET scan done. Polar-maps representing MBF are generated for each rest and stress state using in-house FlowQuant©software. The rest scan will be the baseline. The myocardial blood flow in the four stress scans using hypercapnia as a stress agent will be compared to the rest baseline myocardial blood flow and the adenosine stress scan myocardial blood flow.

SECONDARY OUTCOMES:
Absolute myocardial blood flow differences between end-tidal CO2 scans | Difference between baseline and 60 mmHg PetCO2. Imaging and intervention analysis will be complete in 4 years.
  The effect of increasing doses of pulmonary end-tidal carbon dioxide tension (PetCO2) will be measured and quantification of absolute myocardial blood flow using Rb-82 PET will be calculated. Polar-maps representing MBF are generated for each stress state using in-house FlowQuant©software. Five levels will be measured.
Difference bewteen absolute myocardial blood flow with hypercapnia and with adenosine stress. | Quantification and comparison of the differences in myocardial blood flow with adenosine stress and increasing levels of CO2 as a stress agent. Imaging and intervention analysis will be complete in 4 years.
  The effects of hypercapnia and adenosine on absolute myocardial blood flow using Rb-82 PET will be compared. Polar-maps representing MBF are generated for each stress state using in-house FlowQuant©software.

CONTACTS AND LOCATIONS:
Overall Officials: Terrence D Ruddy, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University Of Ottawa Heart Institute, Ottawa, Ontario, Canada